CLINICAL TRIAL: NCT04469127
Title: This Study is a Phase I/II Clinical Evaluation of a New Investigational Agent, Lutetium-177-DOTAGA-IAC (HurlutinTM Lu-177) to Treat Patients With Unresectable Angiogenic Breast Cancer.
Brief Title: A Phase I/II Multicenter, Open-Label Study of Lu-177-DOTAGA-IAC, for the Treatment of Angiogenic Breast Cancer Patients.
Acronym: Heroine01
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Advanced Imaging Projects, LLC (Industry)
Collaborators: University of Witwatersrand, South Africa (Other); Postgraduate Institute of Medical and Research (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 145358
Record Dates: First submitted 2020-06-30; First posted 2020-07-13 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer Stage IV
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Single Arm study Lu-177-DOTAGA-IAC (intracutaneous)
  Dosage and Dose Escalation Frequency:
  Cohort 1: 75 mCi x 3 (maximum cumulative administered activity, 225mCi) + 100 μgr IAC Cohort 2: 150 mCi x 3 (maximum cumulative administered activity, 450mCi) + 100 μgr IAC Cohort 3: 200 mCi x 3 (maximum cumulative administered activity, 600mCi) + 100 μgr IAC
  Three cycles each 4 weeks apart.
  Interventions: Drug: Lutetium-177-DOTAGA-IAC

INTERVENTIONS:
Drug: Lutetium-177-DOTAGA-IAC — Study participants be administered therapeutic doses of Lutetium-177-DOTAGA-IAC up to three treatments spaced 4 weeks apart.

SUMMARY:
This study is a Phase I/II clinical evaluation of a new investigational agent, Lutetium-177-DOTAGA-IAC (HurlutinTM Lu-177) to treat patients with unresectable angiogenic breast cancer who have previously been treated with at least one prior line of therapy.

DETAILED DESCRIPTION:
This is a prospective, Phase I/II multi-center, interventional open-label study in a total of up to 100 subjects with angiogenic breast cancer. Phase I is to assess the safety and adequacy of a dose of HurlutinTM Lu-177 for up to three cycles, at 4-week intervals. It will include a dose expansion cohort of up to 20 patients. Phase II is to demonstrate the safety, dose adequacy, anti-tumor activity and efficacy of tumor targeted therapy using Lutetium-177-DOTAGA-IAC , as a second- or third-line treatment to extend survival and improve the quality of life of patients with angiogenic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Angiogenic breast tumor by immunohistochemistry confirmation.
2. Positive scan with PET/CT imaging with 18F-FET PET/CT.
3. Tumor progression resistant or refractory to at least one prior lines of standard chemotherapy which include trastuzumab and/or Ado-trastuzumab with or without chemotherapy agents.
4. At least 18 years of age
5. The patient is able and willing to provide informed consent and to comply with the requirements of this trial protocol.
6. ECOG score ≤3
7. Females of childbearing potential must have a negative serum pregnancy test or have had an intervention that renders pregnancy not possible
8. Adequate organ function, defined as:

   1. Absolute neutrophil count (ANC) ≥ 1.5 x 109/mL.
   2. Hemoglobin (Hb) ≥10 g/dl (transfusion or use of EPO is permitted).
   3. Platelets > 100,000/mm3
   4. Creatinine ≤ 1.5 x upper limit of normal (ULN)
   5. AST or ALT ≤ 2.5 x ULN (or ≤5 x ULN in case of liver metastasis)
   6. Alkaline phosphatase ≤2.5 x ULN. Alkaline phosphatase may be more than 2.5 x ULN only in the case of bone metastases, and AST and ALT less than 1.5 x ULN.
   7. Total bilirubin ≤1.5 mg/dl (higher bilirubin levels are permitted if the patient has Gilbert's syndrome).
9. Baseline LVEF ≥40% measured using echocardiogram or equilibrium isotopic ventriculography

Exclusion Criteria:

1. Previously received external beam irradiation that includes more than 30% of bone marrow
2. Previously received external beam irradiation to a field that one kidney.
3. Previously received external beam irradiation to a field that includes the only known lesion.
4. Any uncontrolled significant medical, psychiatric or surgical condition or laboratory finding that would pose a risk to subject safety or interfere with study participation or interpretation of individual subject results.
5. Nephrectomy, renal transplant or concomitant nephrotoxic therapy putting the subject at high risk of renal toxicity during the study.
6. eGFR ≤ 50.
7. Bone metastases are the only known lesions.
8. Patients with a body weight of 400 pounds or more or not able to enter the bore of the PET/CT scanner due to BMI, because of the compromise in image quality with CT, PET/CT and MRI that will result.
9. Inability to lie still for the entire imaging time (e.g., cough, severe arthritis, etc.).
10. Use of any other investigational therapeutic product within 30 days prior to dosing or known requirement for any other investigational agent prior to completion of all scheduled study assessments.
11. Recognized concurrent active infection.
12. Received any live (attenuated) vaccines within 30 days prior to Visit.
13. Recent or chronic treatment with medium-to-high-dose intravenous corticosteroids (methylprednisolone 60 mg/day or hydrocortisone 300 mg/day) within 8 weeks prior to Visit or oral corticosteroids of more than 20 mg prednisone (or equivalent) within 30 days prior to Visit
14. Any unresolved NCI-CTCAE Grade 2 or higher (except alopecia) from previous anti-tumour treatment and/or medical/surgical procedures/interventions.
15. Additional inclusion criterion for measure human dosimetry

    1. Unable to comply with the requirements of the dosimetry imaging protocol
    2. Due to potential radiation safety issues, patients with urinary drainage or diversion (e.g., in-dwelling Foley™ catheter, ureteroileostomy, etc.) will not be enrolled.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-09-30 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Specific Aim 1 | 6 months
  To determine the safety and tolerability of fractionated administrations of 3 cycles of Lu-177-DOTAGA-IAC administered with 4 weeks between cycles in patients with high-risk Angiogenic Breast Cancer who have progressed on, or do not tolerate, best standard-of-care treatment.
  Measurements used to assess the safety, tolerability and side-effects profile will include adverse events of any grade, grade 3 and 4 adverse events, withdrawals due to adverse events and dose reductions due to adverse events. National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE v.5.0) will be used to evaluate AE grade.
Specific Aim 2 | 6 months
  To determine the pharmacokinetics (PK) of Lu-177-DOTAGA-IAC. The area under the Time vs. Concentration curve for Lu-177-DOTAGA-IAC from injection to 72 h
Specific Aim 3 | 6 months
  To determine the whole-body biodistribution of Lu-177-DOTAGA-IAC. Percent injected dose per gram of tissue (%ID)/gm of Lu-177-DOTAGA-IAC.
Specific Aim 4 | 6 months
  To determine the radiation dosimetry of Lu-177-DOTAGA-IAC.Time points will be 0 and 120, 30 and 150, 60 and 180, or 90 and 210 min after injection.Time integrals of activity will be entered into the (Organ Level INternal Dose Assessment/ EXponential Modeling) OLINDA/EXM software.
Specific Aims 5 | 6 months
  To determine optimum cumulative fractionated administered dose. Increase dose range if a DLT (Dose Limiting Toxicity) develops or they do not have a T/B ratio >1.

SECONDARY OUTCOMES:
Specific Aim 1 | 6-12 Months
  To determine the Objective Response Rate (ORR) of fractionated administration of Lu-177-DOTAGA-IAC.Percentage of subjects still alive. Percentage of subjects who achieved a best overall response of Complete Response [CR] or Partial Response [PR] according to RECIST 5.0 Criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Satz, Ph.D., Study Director — Advanced Imaging Projects
Locations (2):
- Postgraduate Institute of Medical and Research, Chandigarh, India
- CM Johannesburg Academic Hospital, University of the Witwatersrand, Johannesburg, South Africa

IPD SHARING:
Plan to Share IPD: Yes
IPD is to be shared with researchers
Supporting Information: CSR
Time Frame: 1 Yr.
Access Criteria: Contact Sponsor

REFERENCES:
- [Result] Baum RP, Kulkarni HR, Muller D, Satz S, Danthi N, Kim YS, Brechbiel MW. First-In-Human Study Demonstrating Tumor-Angiogenesis by PET/CT Imaging with (68)Ga-NODAGA-THERANOST, a High-Affinity Peptidomimetic for alphavbeta3 Integrin Receptor Targeting. Cancer Biother Radiopharm. 2015 May;30(4):152-9. doi: 10.1089/cbr.2014.1747. PMID 25945808
- [Result] Kim YS, Nwe K, Milenic DE, Brechbiel MW, Satz S, Baidoo KE. Synthesis and characterization of alphavbeta(3)-targeting peptidomimetic chelate conjugates for PET and SPECT imaging. Bioorg Med Chem Lett. 2012 Sep 1;22(17):5517-22. doi: 10.1016/j.bmcl.2012.07.024. Epub 2012 Jul 14. PMID 22853992